CLINICAL TRIAL: NCT03328169
Title: Comparative Effectiveness Feasibility Trial for Insomnia Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Hannah Arem, Assistant Professor, George Washington University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121635
Record Dates: First submitted 2017-10-24; First posted 2017-11-01 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer Female; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Active Comparator): Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Mindfulness (Experimental): Mindfulness-Based Therapy
  Interventions: Behavioral: Mindfulness-Based Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Therapy — Participants are taught relaxation and mindfulness techniques to practice. They also learn about various alternative medicine modalities to which they can apply mindfulness with the target of reducing insomnia. The group meets weekly for 2 hours for a duration of 9 weeks.
  Arms: Mindfulness
Behavioral: Cognitive Behavioral Therapy for Insomnia — A licensed psychologist is delivering Cognitive Behavioral Therapy for Insomnia to women for 90-120 minutes weekly for nine weeks. The Cognitive Behavioral Therapy for Insomnia protocol is well documented in published literature.
  Arms: CBT-I

SUMMARY:
Women with breast cancer who report insomnia that started or worsened during breast cancer diagnosis and treatment will be enrolled in a group behavioral trial to one of two arms testing cognitive behavioral therapy for insomnia against a mindfulness-based therapy.

DETAILED DESCRIPTION:
The investigators are recruiting breast cancer survivors with stage I-III or Eastern Cooperative Oncology Group 0-1 breast cancer to enroll in a group-delivered behavioral trial for insomnia. The investigators are comparing mindfulness-based therapies delivered in an alternative medicine context to cognitive behavioral therapy for insomnia. The intervention is 9 weeks, for two hours weekly.

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) Stage I-III or Eastern Cooperative Oncology Group (ECOG) 0-1 breast cancer
* completed active treatment (surgery, radiation, chemotherapy) at least three months prior
* within 5 years of treatment or still on adjuvant therapy
* Completes informed consent to participate

Exclusion Criteria:

* sleep apnea or restless leg syndrome
* practicing mindfulness techniques >1/wk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia | Nine weeks
  Measured using the Insomnia Severity Index (Scale 0-28; higher scores are worse, with 15+ indicating clinical insomnia)
Change in Insomnia | Nine weeks
  Measured using the Pittsburgh Sleep Quality Index (Scale 0-21; higher scores are worse)

SECONDARY OUTCOMES:
Change in cognitive function | Nine weeks
  Measured via the FACT-Cog (Scale 0-132; higher is better)
Change in cognitive function | Nine weeks
  Measured via the Montreal Cognitive Assessment (MOCA)
Change in Fatigue | Nine weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue (Scale 8-40; higher is worse)
Change in Insomnia | Nine weeks
  Measured using an actigraph

CONTACTS AND LOCATIONS:
Locations (1):
- GW Center for Integrative Medicine, Washington D.C., District of Columbia, United States